CLINICAL TRIAL: NCT04709120
Title: Analysis of Health Status of Сomorbid Adult COVID-19 Patients Hospitalised in Second Wave of SARS-CoV-2 Infection
Acronym: ACTIV-2
Status: Completed | Type: Observational
Sponsor: Eurasian Association of Therapists (Other)
Responsible Party: Principal Investigator, Tamara Kriukova, Eurasian Association of Therapists, Eurasian Association of Therapists
Other Study IDs: ACTIV-2
Record Dates: First submitted 2021-01-13; First posted 2021-01-14 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Covid19; Comorbidities and Coexisting Conditions; Risk Factor, Cardiovascular; Death; Diabetes; COPD; Atrial Fibrillation; DVT; CKD
Keywords: Covid19; Comorbidities and Coexisting Conditions; Risk Factor; SARS-CoV-2; COVID-19 Second Wave; COVD-19 First Wave; Death
MeSH Terms: conditions — COVID-19; Death; Diabetes Mellitus; Pulmonary Disease, Chronic Obstructive; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Comparison of COVID-19 disease course in hospitalized patients infected by SARS-CoV-2 in first and second waves of the novel coronavirus infection

DETAILED DESCRIPTION:
Non-commercial depersonalized multi-centered registry study on analysis of chronic non-infectious diseases dynamics after SARS-CoV-2 in first and second waves of the novel coronavirus infection in cohort of Russian adult patients.

Retrospective analysis of medical histories and outcomes in adults with pre-existing conditions after SARS-CoV-2 infection. Comorbidities worsening risk factors measuring through evaluation of range of indicators such as dynamics of diabetes, CKD, COPD, bronchial astma, incidence of hypertonic crises, vascular events and others.

ELIGIBILITY:
Inclusion Criteria:

Suspected or confirmed COVID-19 (according to results of swab-test, antibody test, computed tomography or radiography image)

Exclusion Criteria:

1. Unwillingness to participate in the study;
2. Age under 18.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Anonymized male and female patients over the age of 18 hospitalised since October, 1st, 2020
Sampling Method: Non-Probability Sample
Enrollment: 2968 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
death | 4 weeks
  death for any reason

SECONDARY OUTCOMES:
Number of cases of Acute Kidney Injury depending on Coexisting Conditions | 4 weeks
  Number of cases of Acute Kidney Injury depending on Coexisting Conditions
Number of cases of Myocarditis and Acute Coronary Events depending on Coexisting Conditions | 4 weeks
  Number of cases of Myocarditis and Acute Coronary Events depending on Coexisting Conditions
Number of cases of Cytokine Storm depending on Coexisting Conditions | 4 weeks
  Number of cases of Cytokine Storm depending on Coexisting Conditions
Number of thrombotic and thromboembolic complications of COVID-19 depending on Coexisting Conditions | 4 weeks
  Number of thrombotic and thromboembolic complications of COVID-19 depending on Coexisting Conditions
Decline in GFR excluding Acute Kidney Injury by the time of discharge depending on Coexisting Conditions | 4 weeks
  Decline in GFR excluding Acute Kidney Injury by the time of discharge depending on Coexisting Conditions
Rate of cases of health status worsening occured during hospitalisation | 4 weeks
  Rate of cases of health status worsening occured during hospitalisation

CONTACTS AND LOCATIONS:
Overall Officials: Grigoriy Arutyunov, MD, PhD, Study Director — Eurasian Association of Therapists; Ekaterina Tarlovskaya, MD, PhD, Study Chair — Eurasian Association of Therapists; Aleksander Arutyunov, MD, PhD, Principal Investigator — Eurasian Association of Therapists
Locations (1):
- Eurasian Association of Therapists, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: design of observational studies "Analysis of Chronic Non-infectious Diseases Dynamics After COVID-19 Infection in Adult Patients" and "Analysis of Health Status of Сomorbid Adult COVID-19 Patients Hospitalised in Second Wave of SARS-CoV-2 Infection" — http://russjcardiol.elpub.ru/jour/article/view/4358/
- See also: Lipid profile in hospitalized patients with COVID-19 depending on the outcome of its acute phase: data from the international registry "Dynamics analysis of comorbidities in SARS-CoV-2 infection survivors" — https://russjcardiol.elpub.ru/jour/article/view/5042
- See also: Impact of Kidney Damage on the Course and Prognosis of COVID-19 Infection According to the International Registry "Analysis of Chronic Non-Infectious Diseases Dynamics After Covid-19 Infection in Adult Patients" — https://www.medarhive.ru/jour/article/view/1594/1214
- See also: The impact of carbohydrate metabolism disorders on the early and long-term clinical outcomes of patients with COVID-19 according to the AKTIV and AKTIV 2 registries. — https://www.probl-endojournals.ru/jour/article/view/13175